CLINICAL TRIAL: NCT06694233
Title: Aspirin Prescription For Moderate- and High-Risk Obstetric Population in Outpatient Clnic; A Quality Improvement Project.
Brief Title: Improving Aspirin Prescription Rates in Outpatient Clinic
Status: Terminated | Type: Observational
Why Stopped: Could not obtain ethical approval yet
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Tarek Elkhateb, Dr, Cairo University
Other Study IDs: QIP1
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Low Birth Weight; Small for Gestational Age (SGA); Preeclampsia (PE); Prevention &Amp; Control
Keywords: Aspirin; Preeclampsia; obstetric; risk population
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstetric population candidate for aspirin prescription: Moderate- and high-risk obstetric population
  Interventions: Other: Aspirin prescription on outpatient basis

INTERVENTIONS:
Other: Aspirin prescription on outpatient basis — Improving aspirin prescription rates for candidate patients (moderate- and high-risk obstetric population)

SUMMARY:
Ρrееςlаmpѕia is a syndrome characterised by the new onset of hуреrtеnѕion plus proteinuria, end-organ dysfunction, or both after 20 weeks of gestation. It complicates 3-5% of pregnancies.

Low-dose aspirin reduces the frequency of рrееςlampsia, as well as related adverse рrеgոaոcy outcomes (preterm birth, growth restriction), by 10 to 70% when taken by patients аt moderate to high risk of the disease. It has an excellent maternal/fetal safety profile. Thus, it is a reasonable preventive strategy for these patients.

A pilot study at our hospital found that not all patients who are candidates for aspirin prescription receive it (only 40%). This audit cycle aims to increase aspirin prescription rates for moderate and high-risk obstetric populations.

ELIGIBILITY:
Inclusion Criteria:

Women at high risk are those with any of the following:

1. hypertensive disease during a previous pregnancy
2. chronic kidney disease
3. autoimmune disease such as systemic lupus erythematosus or antiphospholipid syndrome
4. type 1 or type 2 diabetes
5. chronic hypertension.

Women with more than one moderate risk factor, such as are:

1. nulliparity
2. age 40 years or older
3. pregnancy interval of more than 10 years
4. body mass index (BMI) of 35 kg/m2 or more at first visit
5. family history of pre-eclampsia
6. multi-fetal pregnancy.

Exclusion Criteria:

* None. All eligible candidates will be included.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Obstetric population
Study Population: Moderate- and high- risk obstetric population
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Aspirin prescription | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Adan hospital, Al Ahmadi, Al Ahmadi, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh N, Shuman S, Chiofalo J, Cabrera M, Smith A. Missed opportunities in aspirin prescribing for preeclampsia prevention. BMC Pregnancy Childbirth. 2023 Oct 7;23(1):717. doi: 10.1186/s12884-023-06039-w. PMID 37805449
- [Background] Kumar NR, Speedy SE, Song J, Welty LJ, Cavens AD. Quality Improvement Initiative for Aspirin Screening and Prescription Rates for Preeclampsia Prevention in an Outpatient Obstetric Clinic. Am J Perinatol. 2024 May;41(S 01):e917-e921. doi: 10.1055/s-0042-1759705. Epub 2022 Dec 30. PMID 36584691
- See also: Related Info — https://www.nice.org.uk/guidance/cg107

DOCUMENTS (1):
  • Study Protocol (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT06694233/Prot_000.pdf